CLINICAL TRIAL: NCT01203280
Title: Icing Effects on Neck Functions of the Boxers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Physical Education College (Other)
Responsible Party: Shih-Wei Chou, Chang Gung Memorial Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 200800018
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2010-09-16 (Estimated); Status verified 2008-12

CONDITIONS: Balance
Keywords: icing; boxer; balance; neck range of motion; neck isometric strength; balance performance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- balance, neck isometric strength and range of motion (Experimental)
  Interventions: Other: icing massage

INTERVENTIONS:
Other: icing massage — The intervention, ice massage, was conducted by replacing a bag of crushed ice (100 cc) inside a moistened towel and lightly rubbed over lumbosacral region for 10 minutes. The moisture towel increased the intensity of the cooling sensation more than the dry wrappings
  Other Names: serial number:200800018; code name:9700018

SUMMARY:
Most boxing injuries occurs over head and neck which leads to potentially acute or chronic head and neck injuries. Patients with whiplash injury has been reported, reflected by increased body sway and reduced ability to overcome challenging balance tasks. The purpose of this research is to evaluate the fitness and balance outcomes between the boxers and the control group, and boxers undergoing posterior-neck icing effects.

DETAILED DESCRIPTION:
Injuries are common in boxing, occurring most often to the head, neck, face, and hands. Traumatic minor cervical strains are common place in high-impact sports and premature degenerative changes have been documented in sports people exposed to recurrent impact trauma or repetitive forces. Whiplash injury may result in extensive trauma to muscles and ligamentous structures within the cervical spine . Many of these structures, particularly the muscles, contain mechanoreceptors that play a key role in position sense. Studies have shown that head and neck position sense may become impaired following whiplash injury. Subsequently, poor movement patterns, together with the perpetuation of pain and other symptoms may develop.

Posture control is achieved by integration of sensory inputs emanating from somatosensory, vestibular, and visual systems. Patients with whiplash injury has been reported, reflected by increased body sway and reduced ability to overcome challenging balance tasks. In this study we have attempted to evaluate the influence of boxing on balance performances, isometric strength and flexibility; furthermore, evaluate the therapeutic effect of ice massage on boxers.

ELIGIBILITY:
Inclusion Criteria:

* boxers
* Must be able to cooperate to our intervention

Exclusion Criteria:

* Any head and neck injury in recent six months
* personal history of head and neck surgery, tumor, infection, and musculoskeletal disease of neck
* Lesions of central or peripheral nervous system, such as visual or vestibular system, any of which may also affect performance of balance

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2009-01; Primary Completion 2009-04 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
balance performance on the sensory organization test (SOT)

SECONDARY OUTCOMES:
neck isometric strength in six directions
neck range of motion in six directions

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan, Taiwan, Taiwan